CLINICAL TRIAL: NCT06082063
Title: Multifactorial Intervention to Reduce Cardiovascular Disease in Type 1 Diabetes
Acronym: Steno1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Aarhus University Hospital (Other); Steno Diabetes Center Nordjylland (Other); Steno Diabetes Center Odense (Other); Slagelse Hospital (Other); Nykøbing Falster County Hospital (Other); Zealand University Hospital (Other); Hillerod Hospital, Denmark (Other); Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); Regionshospitalet Viborg, Skive (Other); Randers Regional Hospital (Other); Herning Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Regionshospitalet Silkeborg (Other); Bispebjerg Hospital (Other); Regionshospitalet Horsens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNF 22OC0077730
Record Dates: First submitted 2023-05-16; First posted 2023-10-13 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases; Heart Failure; Type 1 Diabetes; Kidney Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Diabetes Mellitus, Type 1; Renal Insufficiency | interventions — Aspirin; semaglutide; (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; finerenone

STUDY DESIGN:
Intervention Model Description: This study uses a PROBE design (prospective, cluster-randomized, open, blinded endpoint evaluation). The study is a superiority trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Multifactorial intervention group (Active Comparator): The multifactorial intervention will be determined by the risk profile and risk markers of each individual and the participants will be allocated to Semaglutide, sotagliflozin or finerenone. The intervention will also comprise more ambitious treatment targets for blood pressure and lipid levels. In addition, all participants will take aspirin 75 mg OD.
  Interventions: Drug: Aspirin tablet; Drug: Semaglutide; Drug: Sotagliflozin; Drug: Finerenone
- Standard intervention group (No Intervention): During the whole study period the standard intervention shall be done according to current Danish and international (ADA/EASD) guidelines. This will address similar risk factors as in the intensive group, but to a less ambitious treatment target for blood pressure and lipid lowering and will not include the use of SGTL2i, finerenone or GLP-1RA, unless these drug classes become recommended in future versions of guidelines.

INTERVENTIONS:
Drug: Aspirin tablet — Antiplatelet treatment: with aspirin 75mg OD is mandatory except for concomitant anticoagulant therapy or allergy. In case of allergy clopidogrel will be used.
  Arms: Multifactorial intervention group
Drug: Semaglutide — GLP-1RA treatment: With semaglutide once weekly individually stepped highest tolerable dose according to standard guidelines aiming at 1 mg/week for persons with HbA1c >53 mmol/mol or BMI>25 kg/m2 and/or ischemic heart disease and/or stroke. For safety see below under benefits and risks. Investigators should pay attention to the need for adjustment in insulin dose after initiation of GLP-1RA treatment.
  Arms: Multifactorial intervention group
Drug: Sotagliflozin — SGLT2i treatment with sotagliflozin 200 mg once daily for persons with UACR >30 mg/g and eGFR < 45 ml/min/1.73 m2 and for persons with a diagnosis of HF. For safety see below under benefits and risks. The limit of eGFR (<45ml/min) for initiation of SGLT2i treatment is set to reduce risk of ketoacidosis. SGLT2i treatment should not be offered to participants on insulin pump therapy, to reduce risk of ketoacidosis. Investigators should pay attention to the need for adjustment in insulin dose after initiation of SGLT2i treatment.
  Arms: Multifactorial intervention group
Drug: Finerenone — Finerenone: 10 mg once daily titrated to 20 mg as add-on in persons with persistent albuminuria (>30 mg/g) despite RAS blockade.
  Arms: Multifactorial intervention group

SUMMARY:
A prospective, randomised, open-labelled, multi-center study. The aim of the Steno 1 study is to test multifactorial intervention in individuals with type 1 diabetes at high risk of CVD with ambitious treatment targets. We will include 2000 participants. Follow-up is 5 years.

DETAILED DESCRIPTION:
Background: Individuals with type 1 diabetes (T1D) are at high risk for cardiovascular disease (CVD). Even with optimal glycemic control, the risk is doubled compared to healthy individuals. Treatment of type 2 diabetes (T2D) is based on multifactorial intervention (MFI). The development of new drug classes has had profound impact on treatment guidelines through a documented reduction in mortality and morbidity in individuals with T2D. MFI acknowledges the need for control and interventions directed towards several risk factors for CVD, and not focus merely on glucose levels. A fundamental change in risk management with a strong focus on MFIs to lower CVD risk in individuals with T1D and comorbidity of CVD, CKD, HF or obesity, has the potential to improve morbidity and survival in T1D.

Objective: The aim of the Steno 1 study is to test MFI in individuals with T1D at high risk of CVD with ambitious treatment targets. We hypothesize, that the MFI reduces major adverse cardiovascular endpoints (MACE) hospitalization for heart failure (HHF), kidney failure and mortality.

Design: This study uses a PROBE design (prospective, cluster-randomized, open, blinded endpoint evaluation), as it will not be possible to mask the MFI. The study is a superiority trial.

Patient population: High-risk individuals with T1D of >10 years duration (>40 years of age with presence of either CKD, CVD, HF, obesity or a >10% 5-year CVD risk determined by the Steno T1 Risk Engine). Participants are recruited from Steno Diabetes Centres or partner clinics.

Randomization: There will be formed three clusters (large patient pool, intermediate- and small). Within each cluster, participating centers will be randomised to either group A or group B. Group A will receive current guideline-recommended standard of care and group B will receive the multifactorial risk based intensive therapy. Participants are allocated to centers based on geography and not based on phenotype.

Intervention: For the intensively treated group, the MFI will be determined by the risk profile and risk markers of each individual and the participants will be allocated to Semaglutide, sotagliflozin, finerenone, ezetimibe and/ or PCSK9-inhibitors. The intervention will also comprise more ambitious treatment targets for blood pressure and lipid levels. In addition, all participants will take aspirin 75 mg OD.

Endpoints: The primary endpoint is to determine whether MFI is superior to standard care with respect to MACE+HHF (composite of time to first non-fatal myocardial infarction, first non-fatal stroke, cardiovascular death or first hospitalization for heart failure). Secondary endpoints are to determine whether MFI is superior to standard care with respect to all-cause mortality, a composite endpoint of renal function (end-stage kidney disease (ESKD) (dialysis, renal death, transplantation) or >50% sustained decline in eGFR) compared to standard of care and to determine whether MFI including the use of SGLT2i and GLP1RA leads to an increased frequency of diabetic ketoacidosis compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Given written informed consent
2. Male or female patients ≥40 years old with type 1 diabetes (diagnosis before age 30 with insulin from onset or if diagnosis after 30 years of age insulin from onset and DKA or positive autoantibodies ( in accordance with local guidelines)) during >10 years.
3. Presence of chronic kidney disease (UACR >30 mg/g or eGFR < 60 ml/min/1.73 m2) OR history of ischemic heart disease (previous myocardial infarction, stroke or angina) OR history of heart failure OR obesity grade 2 and 3 (BMI>35 kg/m2) OR 10-year CVD risk >10% according to Steno Type 1 Risk Engine.
4. Fertile females must use highly efficient chemical, hormonal and mechanical contraceptives during the whole study and at least 2 months after cessation of study drug. The following contraceptive methods are approved: IUD or hormonal contraception that inhibits ovulation, i.e. pills, implantations, transdermal patches, vaginal ring or depot injection. Alternatively, be in menopause (i.e. must not have had regular menstrual bleeding for at least one year), have undergone bilateral oophorectomy or have been surgically sterilized or hysterectomised at least 12 months prior to screening. Fertile participants will be pregnancy tested every six months with urine HCG.
5. Ability to communicate with the investigator and understand informed consent.

Exclusion Criteria:

1. Type 2 diabetes, MODY, secondary diabetes.
2. History of pancreatitis.
3. Body mass index < 18.5 kg/m2
4. Females of childbearing potential who are pregnant, breast-feeding, intend to become pregnant or are not using adequate contraceptive methods.
5. Known or suspected abuse of alcohol or recreational drugs.
6. Participant in another intervention study.
7. CKD stage 5.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
MACE + HHF | 5 years
  Calculate the incidence of cardiovascular events (MACE+HF) to determine whether a multifactorial intervention is superior to standard care with respect to MACE+HHF (composite of time to first non-fatal myocardial infarction, first non-fatal stroke, cardiovascular death or first hospitalization for heart failure).

SECONDARY OUTCOMES:
All-cause mortality | 5 years
  Calculate the incidence of all-cause mortality to determine whether a multifactorial intervention is superior to standard care with respect to all-cause mortality.
Renal function | 5 years
  Calculate the incidence of ESKD to determine whether a multifactorial intervention is superior to standard care with respect to renal function (end-stage kidney disease (ESKD) (dialysis, renal death, transplantation) or >50% sustained decline in eGFR) compared to standard of care.
Diabetic ketoacidosis, safety | 5 years
  Calculate the incidence of DKA to determine whether a multifactorial intervention including the use of SGLT2i and GLP-1RA leads to a change in the frequency of diabetic ketoacidosis compared to standard care.

OTHER OUTCOMES:
Indivudual components of the primary endpoint | 5 years
  To determine whether a multifactorial intervention is superior to standard care with respect to the individual components of the primary endpoint.
Lower extremity amputations | 5 years
  Calculate the incidence of lower extremity amputations to determine whether a multifactorial intervention is superior to standard of care in reducing the total number of lower extremity amputations.
Progression of retinopathy | 5 years
  Calculate the incidence of progression to retinopathy to determine whether a multifactorial intervention is superior to standard of care in reducing progression of retinopathy.
Reduction in kidney function | 5 years
  Calculate the reduction in eGFR (ml/min/1.73m2) to determine whether a multifactorial intervention is superior to standard care with respect to sustained reduction in kidney function (>30% decline in eGFR as well as >40% decline in eGFR).
EQ5D questionnaire | 5 years
  To determine whether a multifactorial intervention is superior to standard care with respect to quality of life as measured with the EQ5D questionnaire.
5- and 10-year cardiovascular risk as assessed using the Steno T1 Risk Engine | 5 years
  To calculate the 5- and 10 year risk of cardiovascular disease at baseline and after 3 and 5 years by the use of the Steno T1 Risk engine to determine whether a multifactorial intervention reduces estimated 5- and 10-year cardiovascular risk compared to standard of care.
Urinary albumin to creatinine ratio (UACR) | 5 years
  Measurement of urinary albumin to creatinine raio (UACR) mg/g at baseline and after 3 and 5 years to determine whether a multifactorial intervention reduces urinary albumin to creatinine ratio (UACR) compared to standard of care.
Decline in eGFR | 5 years
  Measure eGFR (ml/min/1.72 m2) at baseline and after 3 and 5 years to determine whether a multifactorial intervention reduces decline in eGFR compared to standard of care.
HbA1c | 5 years
  Measure HbA1c (mmol/mol) at baseline and after 3 and 5 years to determine whether a multifactorial intervention reduces HbA1c levels compared to standard of care.
LDL cholesteerol | 5 years
  Measure LDL-cholesterol (mmol/L) at baseline and after 3 and 5 years to determine whether a multifactorial intervention reduces LDL cholesterol levels compared to standard of care.
BMI | 5 years
  Measure height (cm) and weight (kg) at baseline and after 3 and 5 years to calculate BMI (kg/m2) to determine whether a multifactorial intervention reduces BMI compared to standard of care.
Biothesiometry | 5 years
  Measure biothesiometry (V) at baseline and efter 3 and years to determine whether a multifactorial intervention reduces biothesiometry score compared to standard of care.
Diabetic ketoacidosis (DKA) | 5 years
  Calculate events of DKA at baeline and after 3 and 5 years to calculate the incidence of DKA to compare incidence of diabetic ketoacidosis between the groups.
Long term risk of CVD events | 10 years
  Calculate the incidence of cardiovascular events (MACE+HHF) at 5 and 10 years to compare in both groups
Survival | 10 years
  Calculate mortality rates after 5 and 10 years to compare overall survival between the groups
Long term risk of ESKD | 10 years
  Calculate rates of ESKD after 5 and 10 years to compare number of individuals developing ESKD in both groups.
Long term risk of lower extremity amputations | 10 years
  Calculate numbers of lower extremity amputations after 5 and 10 years to compare between the groups.
Long term risk of DKA | 10 years
  Calculate the incidence of DKA after 5 and 10 years to compare between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, MD, DMSc, Proffessor, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Steno Diabetes Center Copenhagen, Herlev

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rossing P. Experimental Designs for Multicomponent Interventions in Kidney and Cardiometabolic Diseases. J Am Soc Nephrol. 2024 Oct 1;35(10):1438-1441. doi: 10.1681/ASN.0000000000000449. Epub 2024 Jul 5. No abstract available. PMID 39078403